CLINICAL TRIAL: NCT00809692
Title: In Vivo Functional Assessment of Histamine Pharmacodynamics in Children
Brief Title: In Vivo Assessment of Histamine Pharmacodynamics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn and combined with a new protocol
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10898
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Histamine Biotransformation
Keywords: histamine biotransformation; laser Doppler flowimetry; pediatric pharmacology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 50 subjects with allergic disease receiving histamine challenges by the prick test and iontophoresis technique (serial assessment of blood flow using validated Doppler technique)
  Interventions: Procedure: validated techniques for histamine response
- 2 (Experimental): 150 additional subjects with allergic disease; undergo genotyping; laser Dopper assessment
  Interventions: Procedure: new technique for histamine response

INTERVENTIONS:
Procedure: validated techniques for histamine response — the prick test and iontophoresis technique (serial assessment of blood flow using validated Doppler technique)
  Arms: 1
Procedure: new technique for histamine response — laser Dopper technique and genotyping
  Arms: 2

SUMMARY:
A critical first step to address the "pharmacodynamic information gap" in pediatrics resides with the development of methods capable of accurately measuring the time dependent effects of xenobiotic exposure in a manner sufficient to enable an integrative analysis of drug action which incorporates both pharmacokinetic and pharmacogenetic determinants. The proposed study will evaluate laser Doppler flowimetry, a necessary initial step in developing an "ideal" pharmacodynamic surrogate endpoint that ultimately could be used in infants, children and adolescents to fully characterize the impact of development on the pharmacokinetic (PK) / pharmacodynamic (PD) / pharmacogenetic (PG) determinants of drug effect for agents capable of modulating the cellular response to histamine.

DETAILED DESCRIPTION:
The overall goal of this research is to develop and validate non-invasive approaches suitable for use in pediatrics that are sufficient to directly evaluate genotype-phenotype associations as determinants of the concentration-effect profile of drugs capable of altering microvascular function. The specific goal of this project will be to assess whether microvascular blood flow determined by a previously validated laser Doppler technique can be used as a reliable surrogate endpoint capable of functionally discriminating the effects of polymorphisms in the genes which are quantitatively important for histamine biotransformation. The investigators hypothesize that microvascular blood flow velocity can be used as a valid surrogate marker to discriminate the functional consequences of allelic variants in the enzymes primarily responsible for the biotransformation of histamine.

The project includes two parts:

1. Validation of histamine iontophoresis (with measurement of microvascular blood flow by laser Doppler flowimetry) in a pediatric cohort as a pharmacologic provocation test capable of reliably characterizing the normal physiologic response of the cutaneous microvasculature to this xenobiotic addressed by a study in 50 children with a diagnosis of allergic disease or other "allergic" conditions where treatment with antihistamines represents the medical "standard of care". Subjects will concomitantly (on contralateral extremities) receive histamine challenges by the "gold standard" cutaneous prick test (time dependent response assessed by serial assessment of wheal and flare reactions) and by a previously described iontophoresis technique (time dependent response by serial assessment of microvascular blood flow using a validated laser Doppler technique).Additionally, DNA will be isolated from these subjects for genotyping as described in part 2).
2. Assessment of microvascular response to histamine challenge as a surrogate marker capable of functionally discriminating genotype-phenotype associations for polymorphically expressed genes that are quantitatively important in regulating the biotransformation and pharmacologic inactivation of histamine addressed first by genotyping 150 additional subjects who have an established diagnosis of allergic disease where treatment with antihistamines represents the medical "standard of care". Genotype data for candidate genes of primary interest, histamine-N-methyltransferase (HNMT) and diamine oxidase (DAO), will thus be available from a total of 200 subjects. Based upon known genotype-phenotype associations for HNMT (the enzyme primarily responsible for histamine biotransformation), two cohorts of subjects will be selected from those studied using an extreme discordant phenotype approach: subjects predicted, based upon genotype, to have reduced HMNT activity (i.e., those with 1 or 0 functional alleles) and subjects predicted to have normal enzyme activity (i.e., those with two functional alleles). These study participants will then receive a transcutaneous histamine challenge delivered by iontophoresis, followed by repeated assessment of microvascular reactivity reflected by time-averaged measurement of blood flow velocity using an established laser Doppler technique. Statistical analysis of blood flow velocity and other parameters from the laser Doppler assessment will be used as the primary outcome measurement for comparison of the two study cohorts with respect to expression of HNMT and DAO and the functional consequences thereof, using histamine response as the surrogate assessment of phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between ages of 7 and 18 years
* Diagnosed with allergic disease (i.e., allergic rhinitis, allergic conjunctivitis, allergic asthma)
* Informed consent (Parental permission and subject assent)

Exclusion Criteria:

* Previous history or laboratory evidence of McCune Albright syndrome, immunodeficiency, mastocytosis, receipt of immunomodulatory treatment, chronic conditions associated with abnormalities of the integument, hepatic or renal compromise, neoplastic disease, movement or neurologic disorders and uncontrolled ADHD
* Evidence of atopic dermatitis within a 2 year period from the time of study
* History of previous anaphylactic or anaphylactoid episode
* Evidence of pregnancy (by urinary hCG) or lactation at the time of study
* Receipt of drugs (within a specified time period) of agents capable of altering the response to histamine provocation (e.g., antihistamines, systemic corticosteroids, tricyclic antidepressants)
* Presence of any condition that, in the opinion of the investigator, would produce difficulty with adherence to study procedures.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Statistical analysis of blood flow velocity and other parameters from the laser Doppler assessment | 0

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette L. Jones, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States